CLINICAL TRIAL: NCT05823636
Title: The Clinical Course and Factors for the Progression of Uninvestigated Dyspepsia to Functional Dyspepsia
Status: Recruiting | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, professor, Air Force Military Medical University, China
Other Study IDs: KY20222180-F-5
Record Dates: First submitted 2023-03-26; First posted 2023-04-21 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Dyspepsia
Keywords: Functional Dyspepsia; uninvestigated dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- uninvestigated dyspepsia: Patients aged ≥ 18 years old who had first-onset dyspepsia with one or more symptoms of epigastric pain, epigastric burning, postprandial fullness, early satiation and that has lasted for more than 1 month to 3 months.

SUMMARY:
Dyspepsia is one of the most common gastrointestinal diseases. This disease was defined as predominant epigastric pain lasting for at least 1 month, which can be accompanied with other symptoms, such as epigastric fullness, and early satiety. Despite dyspepsia symptoms lasting for ≥1 month represented clinical problem, a longer duration of 6 months or more after first-onset symptom was required for the diagnosis of functional dyspepsia based on ROME IV criteria. It was unclear about the natural procession of first-onset dyspepsia to functional dyspepsia assessed by Rome IV or Asia criteria and possible factors associated with this progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old who had first-onset dyspepsia with one or more symptoms of epigastric pain, epigastric burning, postprandial fullness, early satiation and that has lasted for more than 1 month to 3 months.

Exclusion Criteria:

1. Patients with local or systemic diseases which may cause dyspeptic symptoms:

   Known active peptic ulcer, cholecystitis, gallstone, gastrointestinal obstruction, gastroparesis, and etc.
2. Known acute or chronic injury of liver or kidney
3. Obvious hematological abnormality, or endocrine and metabolic diseases
4. Known malignancy; Obvious cardiovascular or cerebrovascular diseases (such as coronary heart disease, arrhythmia, cerebral infarction and etc.
5. Other conditions which may be associated with dyspeptic symptoms (such as NSAIDs associated dyspepsia)
6. organ failure defined by Marshall standard or severe psychiatric illnesses
7. pregnancy or lactation
8. unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years old who had first-onset dyspepsia with one or more symptoms of epigastric pain, epigastric burning, postprandial fullness, early satiation and that has lasted for more than 1 month to 3 months.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional dyspepsia defined by ROME IV criteria | 6 months
  Met the following criteria: by one or more of the following symptoms: postprandial fullness, early satiation, epigastric pain, and epigastric burning that are unexplained after a routine clinical evaluation, Criteria fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis.

SECONDARY OUTCOMES:
Functional dyspepsia defined by Asia criteria: | 3 month
  Met the following criteria: by one or more of the following symptoms: postprandial fullness, early satiation, epigastric pain, and epigastric burning that are unexplained after a routine clinical evaluation, the symptoms duration≧3 months.
Global Overall Symptom score (GOSS) | 1month, 3 months, 6 months
  The GOSS consists of 10 cardinal items (epigastric pain, epigastric discomfort, Heartburn, acid regurgitation, upper abdominal bloating, belching, nausea, early satiety, postprandial fullness, other epigastric symptoms(eg. epigastric burning). Each item can be scored from 1 (no) to 7 (worst).
Number of participants subclassified into different subtypes of functional dyspepsia defined by ROME IV criteria | 6 months
  Functional dyspepsia was classified into three subgroups：(1) Postprandial Distress Syndrome, defined as Bothersome postprandial fullness or/and Bothersome early satiation. (2) Bothersome epigastric pain AND/OR Bothersome epigastric burning. (3) mixed syndrome, defined when postprandial distress syndrome and epigastric pain syndrome presented simultaneously.
Short Form of Nepean Dyspepsia Index (SF-NDI) | 1month, 3 months, 6 months
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Hospital anxiety and depression scale | 1month, 3 months, 6 months
  Anxiety and depression of patients are assessed by using Hospital Anxiety and Depression Scale.It contains 14 items (7 anxiety and 7 depression), which assess symptoms experienced during the past week on a 0-3 scale. A subscore of > 8 for depression or anxiety would indicate a clinical case.
Quality of Life scores | 1month, 3 months, 6 months
  Quality of Life scores assessed by Patient-reported outcomes measurement information system (PROMIS) Global-10 questionnaire. PROMIS Global-10 is a newly validated 10-question survey used to assess health care-related quality of life measures for the general population.
  It's a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient and a better quality of life.
Self-reported severity of symptoms by patients | 1 day
  Patients rated the severity of dyspepsia as mild, moderate, and severe by themselves
Number of participants with other functional gastrointestinal diseases defined by ROME IV criteria | 1 day
  Recurrent functional dysphagia， reflux hypersensitivity， irritable bowel syndrome， etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Air Force Military Medical University, China, Xi'an, Shaanxi, China